CLINICAL TRIAL: NCT07138313
Title: Inverkan av Kost pa Dygnsrytmer Och Amnesomsattning
Brief Title: Dietary Impact on Sleep, Rhythms and Related Physiology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CircHFJC2017pt2
Record Dates: First submitted 2025-07-04; First posted 2025-08-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sleep; Diet Interventions; Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: Participants will be studied in a crossover design both after a "healthy diet", and after an "unhealthy diet"
Masking Description: In the crossover condition, participants will not be briefed about what diet they will receive before the actual onset of any of the two dietary interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy diet (Experimental): 'Low-fat dietary intervention' to be administered to participants
  Interventions: Other: Low-fat dietary intervention
- Unhealthier diet (Experimental): 'High-fat dietary intervention' to be administered to participants
  Interventions: Other: High-fat dietary intervention

INTERVENTIONS:
Other: Low-fat dietary intervention — Low-fat diet for approximately 1 week, preceding in-lab study period (approximately 2 days) under standardized conditions (total dietary exposure up to 9-10 days).
  Arms: Healthy diet
Other: High-fat dietary intervention — High-fat diet for approximately 1 week, preceding in-lab study period (approximately 2 days) under standardized conditions (total dietary exposure up to 9-10 days).
  Arms: Unhealthier diet

SUMMARY:
Sleep and metabolism are closely interconnected, and emerging evidence suggests that dietary composition may influence both sleep quality and key physiological functions such as glucose regulation, cardiovascular activity, and hormonal signaling. This study aims to investigate how a Western-style unhealthy diet versus a healthier, fiber-rich diet affects objective and subjective sleep measures, 24-hour physiological parameters, and a range of biomarkers related to cardiometabolic, neurodegenerative, and gut microbial function.

DETAILED DESCRIPTION:
Metabolism is tightly regulated by sleep and interacts bidirectionally with diet. While it is well established that insufficient or disrupted sleep can impair glucose regulation, cardiovascular function, and promote unhealthy eating behaviors that promote cardiometabolic disease, less is known about how different dietary patterns impact subjective and objective sleep parameters, as well as related physiological systems.

The study will systematically investigate how consumption of an unhealthier "Western" diet, compared to a healthier diet, affects both objective and subjective sleep parameters, as well as 24-hour heart rate and blood pressure profiles, glucose variability, and hormonal and molecular biomarkers.

The study will be conducted as a 2-condition, randomized crossover study, with assessments in the field for about a week, followed by a multi-day stay for measurements under standardized laboratory conditions. Participants will be monitored using polysomnography, and wearable devices, including for continuous glucose and heart rate parameters, with multi-compartment sampling to assess diet-mediated responses across cardiometabolic, neurodegenerative, and microbial pathways. In field and in the lab, biological samples will be collected repeatedly across the day to establish diurnal rhythms.

Cognitive performance, mood, and subjective appetite will also be evaluated. By identifying diet-driven changes in sleep and related physiological functions, this study aims to provide mechanistic insights into how nutrition impacts sleep, cardiometabolic health parameters and molecular pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-32 yr
* Healthy (self-reported) and not on chronic medication
* BMI 18-27 kg/m2 (and waist circumference <102 cm), and weight stable (less than 5% body weight change in the past 6 months)
* Non-smoker and non-nicotine user
* Regular sleep-wake pattern, with sleep duration of 7-9.25 hrs per night
* Regular exercise habits the last 2 months
* Regular daily meal pattern with 3 main meals

Exclusion Criteria:

* Major or chronic illness, e.g. diabetes, renal disease or inflammatory bowel disease
* Current or history of endocrine or metabolic disorders
* Psychiatric or neurological disorders (e.g. bipolar disorder, epilepsy)
* Frequent gastrointestinal symptoms
* Chronic medication
* Any sleep disorder (including recent or chronic symptoms of insomnia)
* Shift work in the preceding three months or for a long duration
* Extreme chronotype or physical activity patterns
* Time travel over two time zones in the preceding month
* Too much weight gain or weight loss in the preceding 6 months (±5% body weight in past 6 months)
* Any issues with or allergies against the provided food items
* Recent major dietary changes or adoption of specific dietary regimens
* Women who are pregnant, breastfeeding, or planning to become pregnant during the study period.
* Use of illicit drugs or substances of abuse

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Architecture and Neurophysiological Features | Up to 9 nights on each diet
  Objective registration and analysis of sleep, based on polysomnography or validated wearable devices to capture macrosleep, spectral and microsleep features.
Change in 24-Hour Heart Rate Variability (HRV) | Up to 9 days on each diet
  Continuous measurement of HRV, using a wearable device, focused on the metric Root Mean Square of the Successive Differences (RMSD); additional metrics (Standard Deviation of NN intervals (SDNN), low frequency to high frequency (LF/HF) ratio) analyzed for exploratory purposes.

SECONDARY OUTCOMES:
24-Hour Heart Rate (HR) | Up to 9 days on each diet
  Continuous measurement of heart rate using a wearable device
Heart Rate Response to Standardized Stair Stepping | Baseline and day 7-9 of each diet period
  ECG-based heart rate measured at baseline, during stepping and repeatedly (up to 5 min) post-stair stepping, to assess recovery, also analyzed in relation to sleep metrics.
Morning-to-Evening and 24-h blood pressure (BP) | Up to 9 days on each diet
  Morning, evening, and 24-h ambulatory measurement of systolic blood pressure, also analyzed in relation to sleep metrics.
24 Hour Continuous Glucose Levels | Up to 9 days on each diet
  Continuous (24-h) monitoring of interstitial glucose for analysis of mean levels and variability metrics (e.g., SD, coefficient of variation, postprandial changes), also analyzed in relation to sleep metrics.
Levels of Blood-based Biomarkers | Up to 9 days on each diet
  Changes in levels of molecular factors such as DNA, hormones/proteins and metabolites, due to the preceding dietary intervention, and also in relation to sleep metrics.
Levels of CNS biomarkers | Up to 9 days on each diet
  Levels of CNS health biomarkers (such as brain-derived neurotrophic factor (BDNF), Tau (e.g. BD-tau) and Amyloid beta (Aβ) species, glial fibrillary acidic protein (GFAP), and Neurofilament light chain (NfL)).
Urinary Metabolite Levels | Up to 9 days on each diet
  Urine levels of excretion molecules (such as melatonin breakdown metabolites).
Change in Metabolic Fuel Utilization | Up to 9 days on each diet
  Change in metabolic fuel utilization as measured by respirometry, in response to the dietary interventions.
Levels of Fecal Metabolites | Up to 9 days on each diet
  Changes in levels of fecal metabolites (such as short chain fatty acids, bile acids) due to each dietary intervention
Levels of Fecal Microbiota | Up to 9 days on each diet
  Changes in fecal microbiota (metagenomic, compositional) due to each dietary intervention
Levels of Salival Biomarkers | Up to 9 days on each diet
  Changes in levels of salival molecules (such as cortisol and melatonin), also in relation to sleep-circadian metrics.
Levels of Salival Microbiota | Up to 9 days on each diet
  Changes in salival microbiota (metagenomic, compositional) due to each dietary intervention
Changes in glucose tolerance | Day 8-9 on each diet
  Glucometabolic response to a standardized 2-h glucose tolerance test, also analyzed in relation to sleep-circadian metrics.
Levels of Immune Cells | Up to 9 days on each diet
  Immune cell profile across the day in response to each diet
Change in Subjective Sleep Quality | Up to 9 days on each diet
  Change in self-reported sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI), supplementing objective sleep data. Total Score (0-21; higher = worse).
Subjective Hunger and Appetite Levels | Up to 9 days on each diet
  Self-reported hunger and appetite across the day, and prior to and after meals, as assessed via visual analogue scales (VAS, i.e., with scores 0 for the lowest subjective rating, to 100 for the highest rating)
Body Temperature | Up to 9 days on each diet
  Body temperature measured via wearable sensors to assess effects of dietary interventions on thermoregulation and its relationship to sleep, circadian rhythms and metabolism.
Change in Composite Cognitive Performance Score | Up to 9 days on each diet
  Composite score from four tasks:
  1. Psychomotor Vigilance Task (PVT) - sustained attention; faster reaction times and fewer lapses corresponds to better performance;
  2. Go/No-Go Task - inhibitory control; higher accuracy on no-go trials and faster correct go responses corresponds to better performance;
  3. Task-Switching Task - cognitive flexibility; smaller switch cost (difference in reaction time between switch and repeat trials) and higher accuracy corresponds to better performance;
  4. Memorability Task - episodic memory; higher hit rate (0-100%) and fewer false alarms corresponds to better performance.
  All scores will be standardized and averaged; higher composite values indicate better cognitive performance.
Changes in mental wellbeing | Up to 9 days on each diet
  Self-reported assessment of mental wellbeing using validated subjective scales (visual analogue scales going from lowest 0 to highest of 100), to evaluate effects of diet and sleep.
Changes in Central Hemodynamics | Up to 9 days on each diet
  Morning, evening, and 24-h ambulatory levels of central hemodynamics reflecting central blood pressure and arterial resistance, also analyzed in relation to sleep metrics
Effect Modification by Biological Sex | Based on data collected up to 9 days on each diet
  Exploratory subgroup analysis to determine if male vs. female participants differ in response to dietary interventions, for primary and secondary outcomes
Effect Modification by Cardiorespiratory Fitness | Based on data collected up to 9 days on each diet
  Exploratory analysis to determine whether cardiorespiratory fitness parameters modulates responses to how the diets impact primary and secondary outcomes.
Change in Dim Light Melatonin Onset | Up to 9 days on each diet
  Dim Light Melatonin Onset as assessed via repeatedly measured melatonin levels, measured in the evening under standardized conditions
Levels of molecular biomarkers in dried blood spots | Up to 9 days on each diet
  Analysis of levels of molecular biomarkers (such as CRP) in dried blood spots from finger samples, and how these correlate with biomarker levels from peripheral venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cedernaes, MD, PhD, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Uppsala biomedical center, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No